CLINICAL TRIAL: NCT05937126
Title: Rapid Diagnostic Supporting Antimicrobial Stewardship in Patients With Pneumonia (RASP) - A Quality Improvement Theragnostic Stewardship Project
Brief Title: Rapid Diagnostic Supporting Antimicrobial Stewardship in Patients With Pneumonia
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robin Patel, Principal Investigator, Mayo Clinic
Other Study IDs: 19-012521
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Lower Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard culture and antimicrobial susceptibility testing (AST): Lower respiratory tract sputum samples (expectorated sputum, induced sputum, tracheal secretions, or bronchoalveolar lavage) collected in the inpatient setting per standard of care from adults with lower respiratory tract infections will receive standard culture and antimicrobial susceptibility testing (AST).
  Interventions: Diagnostic Test: Culture and antimicrobial susceptibility testing
- Standard culture and AST PLUS rapid identification and AST: Lower respiratory tract sputum samples (expectorated sputum, induced sputum, tracheal secretions, or bronchoalveolar lavage) collected in the inpatient setting per standard of care from adults with lower respiratory tract infections will receive standard culture and AST PLUS rapid identification and AST using the FDA-approved/cleared FilmArray Pneumonia Panel
  Interventions: Diagnostic Test: FilmArray Pneumonia Panel; Diagnostic Test: Culture and antimicrobial susceptibility testing

INTERVENTIONS:
Diagnostic Test: FilmArray Pneumonia Panel — FDA-approved/cleared molecular, multiplex device that rapidly identifies viruses, bacteria, and antimicrobial resistance genes in sputum-like and bronchoalveolar lavage (BAL)-like specimens obtained from individuals with signs of a lower respiratory tract infection.
  Groups: Standard culture and AST PLUS rapid identification and AST
Diagnostic Test: Culture and antimicrobial susceptibility testing — Standard of care Gram stain, culture and other clinically ordered tests will be performed per standard practice.

SUMMARY:
The purpose of this study is to determine whether or not the FilmArray Penumonia Panel adds value to patient care.

ELIGIBILITY:
Inclusion Criteria:

- Subjects who have the following samples collected and submitted for culture as part of routine clinical practice: Expectorated sputum, induced sputum, tracheal secretions, bronchoalveolar lavage.

Exclusion Criteria:

* Subjects who do not have MN Research Authorization on file
* Rejected sputum culture (i.e., due to low quality)
* Positive respiratory cultures within prior 7 days
* Deceased at time of sample randomization
* Any subject affected by Global Data protection Regulation (GDPR)
* Previous enrollment in the study.
* Outpatient status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lower respirator tract samples obtained from inpatient settings only (medical/surgical floors and intensive care units) at Mayo Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 1203 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Time until first modification of antibiotic therapy | 96 hours
  Mean time until first modification of antibiotic therapy (in hours)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Patel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Virk A, Strasburg AP, Kies KD, Donadio AD, Mandrekar J, Harmsen WS, Stevens RW, Estes LL, Tande AJ, Challener DW, Osmon DR, Fida M, Vergidis P, Suh GA, Wilson JW, Rajapakse NS, Borah BJ, Dholakia R, Reed KA, Hines LM, Schuetz AN, Patel R. Rapid multiplex PCR panel for pneumonia in hospitalised patients with suspected pneumonia in the USA: a single-centre, open-label, pragmatic, randomised controlled trial. Lancet Microbe. 2024 Dec;5(12):100928. doi: 10.1016/S2666-5247(24)00170-8. Epub 2024 Oct 17. PMID 39426396
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials